CLINICAL TRIAL: NCT05827185
Title: Combined and Isolated Effects of Workstation Ergonomics and Physiotherapy in Improving Cervicogenic Headache and Work Ability in Office Workers - A Single-blinded, Randomized Controlled Study.
Brief Title: Effects of Workstation Ergonomics and Physiotherapy in Cervicogenic Headache.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prince Sattam Bin Abdulaziz University (Other)
Responsible Party: Principal Investigator, Gopal Nambi, Associate Professor, Prince Sattam Bin Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: RHPT/019/082
Record Dates: First submitted 2023-04-12; First posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Cervicogenic Headache
Keywords: Workstation; Ergonomics; Physiotherapy; Randomized control trial; Office workers
MeSH Terms: conditions — Post-Traumatic Headache | interventions — Physical Therapy Modalities; Patient Education as Topic

STUDY DESIGN:
Intervention Model Description: The study includes ergonomic modifications group (EMG; n=24), physiotherapy group (PTG; n=24), and ergonomic modifications combined with physiotherapy group (EPG; n=24) and, control group (CNG; n=24)
Who Masked: Outcomes Assessor
Masking Description: Because of the experimental nature of the study methodology, it was not feasible to blind the treating therapist as well as the participants included in the study. The therapists who assessed the outcome variables at baseline, 4-weeks, 8-weeks, and 6-months were blinded. Therefore, the therapist providing the treatment and the therapist measuring the data were different individuals. In addition, the outcome-measuring therapist continued to be masked to the participant's groups at all-time intervals. Also, participants were asked not to discuss their treatment details with their peers or the outcome-measuring therapist.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Ergonomic modifications group (EMG) (Experimental): A blinded therapist used an observation-based ergonomics assessment check list for office workers to check the status of office environment, which usually took 40 - 45 minutes to complete. It consists of 5 domains. After assessment required modifications were done in the chair, desk, keyboard, mouse, computer screen, telephone and the office environment. Ergonomic education and instructions were also given on an individual basis as per the report of the assessment.
  Interventions: Biological: Ergonomic modifications
- Physiotherapy group (PTG) (Experimental): First of all, hydro collator pack was applied over the neck region for 10 minutes to relax the muscles of the neck region. Then the therapist located the sites of abnormal changes in each vertebra and then cervical manipulation was given. If any participant reported any new red flag signs or showed no signs for manipulation, such as no pain or musculoskeletal dysfunction, then the procedure was not performed.
  Interventions: Biological: Physiotherapy
- Ergonomic modifications combined with physiotherapy group (EPG) (Experimental): A blinded therapist used an observation-based ergonomics assessment check list for office workers to check the status of office environment, which usually took 40 - 45 minutes to complete. It consists of 5 domains. After assessment required modifications were done in the chair, desk, keyboard, mouse, computer screen, telephone and the office environment. Ergonomic education and instructions were also given on an individual basis as per the report of the assessment.
  First of all, hydro collator pack was applied over the neck region for 10 minutes to relax the muscles of the neck region. Then the therapist located the sites of abnormal changes in each vertebra and then cervical manipulation was given. If any participant reported any new red flag signs or showed no signs for manipulation, such as no pain or musculoskeletal dysfunction, then the procedure was not performed.
  Interventions: Biological: Ergonomic modifications and Physiotherapy
- Control group (CNG) (Sham Comparator): Participants in the CNG group received the patient education through an experienced physiotherapist and each session lasting for 30 minutes for 4 weeks. According to each individual patients' abilities the therapist educated them to improve the health literacy regarding the condition. The therapist educated them about the benefits of self-care activities, maintaining good posture, stay active and doing active movements and stretching muscles for preventing the health related musculoskeletal injuries at the workstation. Also, life style modifications were taught to the patients to prevent further deterioration of the condition.
  Interventions: Biological: Patient education

INTERVENTIONS:
Biological: Ergonomic modifications — A blinded therapist used an observation-based ergonomics assessment check list for office workers to check the status of office environment, which usually took 40 - 45 minutes to complete. It consists of 5 domains (7 items related to office chair, 9 items related to office desk, 8 items related to keyboard and mouse, 5 items related to computer screen, 3 items related to telephone and 5 items related to the office environment -) and it has a good reliability and validity. After assessment required modifications were done in the chair, desk, keyboard, mouse, computer screen, telephone and the office environment. Ergonomic education and instructions were also given on an individual basis as per the report of the assessment.
  Arms: Ergonomic modifications group (EMG)
Biological: Physiotherapy — First of all, hydro collator pack was applied over the neck region for 10 minutes to relax the muscles of the neck region. Then the therapist located the sites of abnormal changes in each vertebra and then cervical manipulation was given. To perform the C1-C2 cervical spine manipulation (CSM) the participant was instructed to lie in a face-up position with upper and lower extremities kept aside relaxed. The head was kept in a neutral position and the treating therapist stands at the patient's head side and holds the chin of the patient with the right side hand. The therapist left hand holds the posterior aspect of the head and does two to three free rotatory movements. Afterwards, the therapist did HVLAT technique in either the right or left direction based upon the symptoms informed by the patient.
  Arms: Physiotherapy group (PTG)
Biological: Ergonomic modifications and Physiotherapy — A blinded therapist used an observation-based ergonomics assessment check list for office workers to check the status of office environment, which usually took 40 - 45 minutes to complete. After assessment required modifications were done in the chair, desk, keyboard, mouse, computer screen, telephone and the office environment.
  First of all, hydro collator pack was applied over the neck region for 10 minutes to relax the muscles of the neck region. Then the therapist located the sites of abnormal changes in each vertebra and then cervical manipulation was given.
  Arms: Ergonomic modifications combined with physiotherapy group (EPG)
Biological: Patient education — Participants in the CNG group received the patient education through an experienced physiotherapist and each session lasting for 30 minutes for 4 weeks. According to each individual patients' abilities the therapist educated them to improve the health literacy regarding the condition. The therapist educated them about the benefits of self-care activities, maintaining good posture, stay active and doing active movements and stretching muscles for preventing the health related musculoskeletal injuries at the workstation. Also, life style modifications were taught to the patients to prevent further deterioration of the condition.
  Arms: Control group (CNG)

SUMMARY:
Cervicogenic headache (CgH) is a distinct form of headache and accounts for 17.8% of all headaches and the prevalence rate is between 0.4% and 20%. A guide to health and safety in the office handbook by common wealth of Australia (2008) suggested the ergonomic guidance and interventions for preventing and treating musculoskeletal disorder (MSD) injuries in the office workers. Also, It has been estimated that 34% of US citizens receive some sort of physiotherapy for CgH each year. However, no studies have compared and investigated the combined and individual effects of workstation ergonomics, physiotherapy and patient education for improving cervicogenic headache and work ability in office workers.

DETAILED DESCRIPTION:
Cervicogenic headache (CgH) is a distinct form of headache and accounts for 17.8% of all headaches and the prevalence rate is between 0.4% and 20%. A guide to health and safety in the office handbook by common wealth of Australia (2008) suggested the ergonomic guidance and interventions for preventing and treating musculoskeletal disorder (MSD) injuries in the office workers. Also, It has been estimated that 34% of US citizens receive some sort of physiotherapy for CgH each year. However, no studies have compared and investigated the combined and individual effects of workstation ergonomics, physiotherapy and patient education for improving cervicogenic headache and work ability in office workers.

Therefore, our study objective was intended to compare and investigate the combined and individual effects of workstation ergonomics, physiotherapy and patient education in improving cervicogenic headache and work ability in office workers. This randomized clinical trial hypothesized that there is a difference in primary and secondary outcome measures between workstation ergonomics, physiotherapy and patient education for improving cervicogenic headache and work ability in office workers.

ELIGIBILITY:
Inclusion Criteria:

Patients aged between 18-60 years Working in the computer ≥ 32 hrs/week Suffering from Cervicogenic Headache (>3 months) Pain intensity ≥3 on a numerical pain rating scale (NPRS), Cervicogenic Headache resulting from pain in the neck followed by headache, Limited neck movements, Neck muscle spasm, Consent to participate in the study

Exclusion Criteria:

Other primary headaches such as migraine and tension-type headaches (TTH), Whiplash injuries, Participants who show signs of the five 'D's' (dizziness, drop attacks, dysarthria, dysphagia, diplopia) Who have signs of the three 'N's (nystagmus, nausea, other neurological symptoms (cord compression or nerve root involvement), Contraindications to physio therapy (Congenital anomalies, tumor, degenerative and inflammatory arthritis, osteoporosis, dislocation, fractures, and steroid intake), Underwent previous head and neck surgeries, Had physiotherapy or other complementary therapies in the last three months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
CgH frequency | Baseline
  It is a self-administered outcome variable where the patient enters his CgH pain experience in a medical log book every evening to find the number of painful days in 4-weeks
CgH frequency | 4 weeks
  It is a self-administered outcome variable where the patient enters his CgH pain experience in a medical log book every evening to find the number of painful days in 4-weeks
CgH frequency | 8 weeks
  It is a self-administered outcome variable where the patient enters his CgH pain experience in a medical log book every evening to find the number of painful days in 4-weeks
CgH frequency | 6 months
  It is a self-administered outcome variable where the patient enters his CgH pain experience in a medical log book every evening to find the number of painful days in 4-weeks

SECONDARY OUTCOMES:
CgH pain intensity | Baseline
  The pain intensity of CgH was assessed using an 11-point numerical pain rating scale (NPRS). Patients rated their typical level of pain status during the previous week on a 10 cm horizontal line, with one end 0 representing "no pain" and the other end 10 representing "worst pain imaginable.
CgH pain intensity | 4 weeks
  The pain intensity of CgH was assessed using an 11-point numerical pain rating scale (NPRS). Patients rated their typical level of pain status during the previous week on a 10 cm horizontal line, with one end 0 representing "no pain" and the other end 10 representing "worst pain imaginable.
CgH pain intensity | 8 weeks
  The pain intensity of CgH was assessed using an 11-point numerical pain rating scale (NPRS). Patients rated their typical level of pain status during the previous week on a 10 cm horizontal line, with one end 0 representing "no pain" and the other end 10 representing "worst pain imaginable.
CgH pain intensity | 6 months
  The pain intensity of CgH was assessed using an 11-point numerical pain rating scale (NPRS). Patients rated their typical level of pain status during the previous week on a 10 cm horizontal line, with one end 0 representing "no pain" and the other end 10 representing "worst pain imaginable.
CgH disability | Baseline
  The Headache Impact Test (HIT) questionnaire is a valid and reliable instrument to assess the level of disability in CgH patients. It consists of six items: pain, social functioning, role functioning, vitality, cognitive functioning, and psychological distress. The score categories are no or mild disability (49 or less), moderate disability (50-55), severe disability (56-59), and complete disability (60-78).
CgH disability | 4 weeks
  The Headache Impact Test (HIT) questionnaire is a valid and reliable instrument to assess the level of disability in CgH patients. It consists of six items: pain, social functioning, role functioning, vitality, cognitive functioning, and psychological distress. The score categories are no or mild disability (49 or less), moderate disability (50-55), severe disability (56-59), and complete disability (60-78).
CgH disability | 8 weeks
  The Headache Impact Test (HIT) questionnaire is a valid and reliable instrument to assess the level of disability in CgH patients. It consists of six items: pain, social functioning, role functioning, vitality, cognitive functioning, and psychological distress. The score categories are no or mild disability (49 or less), moderate disability (50-55), severe disability (56-59), and complete disability (60-78).
CgH disability | 6 months
  The Headache Impact Test (HIT) questionnaire is a valid and reliable instrument to assess the level of disability in CgH patients. It consists of six items: pain, social functioning, role functioning, vitality, cognitive functioning, and psychological distress. The score categories are no or mild disability (49 or less), moderate disability (50-55), severe disability (56-59), and complete disability (60-78).
Cervical flexion-rotation test (FRT) | Baseline
  The cervical flexion-rotation test is done with the patient in a supine lying position. The therapist passively maintains the patient's neck into full flexion to relax the structures of the middle and lower cervical spine, then the patient's head is passively rotated in each direction while the flexed position is maintained and the range of motion is measured.
Cervical flexion-rotation test (FRT) | 4 weeks
  The cervical flexion-rotation test is done with the patient in a supine lying position. The therapist passively maintains the patient's neck into full flexion to relax the structures of the middle and lower cervical spine, then the patient's head is passively rotated in each direction while the flexed position is maintained and the range of motion is measured.
Cervical flexion-rotation test (FRT) | 8 weeks
  The cervical flexion-rotation test is done with the patient in a supine lying position. The therapist passively maintains the patient's neck into full flexion to relax the structures of the middle and lower cervical spine, then the patient's head is passively rotated in each direction while the flexed position is maintained and the range of motion is measured.
Cervical flexion-rotation test (FRT) | 6 months
  The cervical flexion-rotation test is done with the patient in a supine lying position. The therapist passively maintains the patient's neck into full flexion to relax the structures of the middle and lower cervical spine, then the patient's head is passively rotated in each direction while the flexed position is maintained and the range of motion is measured.
Work ability | Baseline
  It was measured by Work Ability Index (WAI), which consists of 7 items such as: current ability, work ability in relation to physical and mental demands of the job, reported diagnosed diseases, estimated impairment due to health status, sick leave over the last 12 months, self-prognosis of work ability in the 2 years to come and mental resources of the individual. It ranges from 7 to 49 points and 4 categories such as; poor (7 - 27), moderate (28 -36), good (37-43) and excellent (44-49).
Work ability | 4 weeks
  It was measured by Work Ability Index (WAI), which consists of 7 items such as: current ability, work ability in relation to physical and mental demands of the job, reported diagnosed diseases, estimated impairment due to health status, sick leave over the last 12 months, self-prognosis of work ability in the 2 years to come and mental resources of the individual. It ranges from 7 to 49 points and 4 categories such as; poor (7 - 27), moderate (28 -36), good (37-43) and excellent (44-49).
Work ability | 8 weeks
  It was measured by Work Ability Index (WAI), which consists of 7 items such as: current ability, work ability in relation to physical and mental demands of the job, reported diagnosed diseases, estimated impairment due to health status, sick leave over the last 12 months, self-prognosis of work ability in the 2 years to come and mental resources of the individual. It ranges from 7 to 49 points and 4 categories such as; poor (7 - 27), moderate (28 -36), good (37-43) and excellent (44-49).
Work ability | 6 months
  It was measured by Work Ability Index (WAI), which consists of 7 items such as: current ability, work ability in relation to physical and mental demands of the job, reported diagnosed diseases, estimated impairment due to health status, sick leave over the last 12 months, self-prognosis of work ability in the 2 years to come and mental resources of the individual. It ranges from 7 to 49 points and 4 categories such as; poor (7 - 27), moderate (28 -36), good (37-43) and excellent (44-49).

CONTACTS AND LOCATIONS:
Overall Officials: Gopal Nambi, PhD, Principal Investigator — Prince Sattam bin Abdulaziz University, Al Kharj, Saudi Arabia
Locations (1):
- Dr. Gopal Nambi, Al Kharj, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
The data can be obtained through contacting the corresponding author.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within one week

REFERENCES:
- [Derived] Nambi G, Alghadier M, Pakkir Mohamed SH, Vellaiyan A, Ebrahim EE, Sobeh DE, Kashoo FZ, Albarakati AJA, Alshahrani NA, Eswaramoorthi V. Combined and isolated effects of workstation ergonomics and physiotherapy in improving cervicogenic headache and work ability in office workers: a single-blinded, randomized controlled study. Front Public Health. 2024 Nov 28;12:1438591. doi: 10.3389/fpubh.2024.1438591. eCollection 2024. PMID 39697289